CLINICAL TRIAL: NCT01829334
Title: A Comparative Study on the Cost-effectiveness of Four Methods in Preventing Fissure Caries in Permanent Teeth
Brief Title: Cost-effectiveness of Four Methods in Preventing Fissure Caries in Permanent Teeth
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, LO, Edward Chin Man, Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: UW 06-203
Record Dates: First submitted 2013-04-08; First posted 2013-04-11 (Estimated); Last update posted 2013-04-11 (Estimated); Status verified 2013-04

CONDITIONS: Dental Caries
Keywords: dental caries
MeSH Terms: conditions — Dental Caries | interventions — Bifluorid 12

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Resin dental sealant (Active Comparator): Resin dental sealant placed on pits and fissures of first permanent molars, single-time placement and no replacement
  Interventions: Other: Resin dental sealant
- ART dental sealant (Experimental): ART dental sealant placed with glass ionomer material using the ART technique on permanent first molar, single-time placement and no replacement
  Interventions: Other: ART dental sealant
- Sodium fluoride varnish (Experimental): Topical application of 5% sodium fluoride varnish onto pits and fissures of permanent first molars, repeated every 6 months
  Interventions: Other: Sodium fluoride varnish
- Silver fluoride solution (Experimental): Topical application of 38% silver fluoride solution onto pits and fissures of permanent first molars, repeated every 12 months
  Interventions: Other: Silver fluoride solution

INTERVENTIONS:
Other: ART dental sealant — ART dental sealant placed with glass ionomer material using the ART technique on permanent first molar, single-time placement and no replacement
  Arms: ART dental sealant
Other: Resin dental sealant — Resin dental sealant placed on pits and fissures of first permanent molars, single-time placement and no replacement
  Arms: Resin dental sealant
Other: Sodium fluoride varnish — Topical application of 5% sodium fluoride varnish onto pits and fissures of permanent first molars, repeated every 6 months
  Arms: Sodium fluoride varnish
Other: Silver fluoride solution — Topical application of 38% silver fluoride solution onto pits and fissures of permanent first molars, repeated every 12 months
  Arms: Silver fluoride solution

SUMMARY:
The aim of this proposed study is to investigate the cost-effectiveness of four methods in preventing fissure caries in permanent teeth, which is the most prevalent dental disease in primary school children in China.

The four caries prevention methods are: resin fissure sealant, atraumatic restorative treatment (ART) sealant, sodium fluoride varnish, and silver diamine fluoride (SDF) solution.

The specific study objectives are:

1. to describe longitudinally the clinical outcomes of using the above four methods to prevent dental caries in the pits and fissures of permanent first molars in school children,
2. to describe the cost of using the above four methods to prevent dental caries in an outreaching dental care programme in China, and
3. to compare the cost-effectiveness of the above four caries prevention methods.

ELIGIBILITY:
Inclusion Criteria:

* school children in good general health
* has at least one pair of sound permanent first molars with deep occlusal fissures or fissures with signs of early caries

Exclusion Criteria:

* children with major systemic disease or on long-term medication
* children not cooperative and refuse dental treatments

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 329 (Actual)
Dates: Start 2006-06; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
dental caries | 3 years
  development of carious cavity after 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Edward CM Lo, Principal Investigator — The University of Hong Kong
Locations (1):
- Primary schools, Shenzhen, China

REFERENCES:
- [Derived] Liu BY, Xiao Y, Chu CH, Lo EC. Glass ionomer ART sealant and fluoride-releasing resin sealant in fissure caries prevention--results from a randomized clinical trial. BMC Oral Health. 2014 May 19;14:54. doi: 10.1186/1472-6831-14-54. PMID 24886444